CLINICAL TRIAL: NCT00802165
Title: Effect of Electroacupuncture on Pain Threshold
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. John Zhang, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR0806080149
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Pain
Keywords: Asymptomatic normals
MeSH Terms: conditions — Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture Treatment Group (Experimental): Group is given a total of four electroacupuncture treatments to evaluate it's anesthetic effectiveness
  Interventions: Device: Electroacupuncture
- Sham Treatment Group (Sham Comparator): Sham electroacupuncture treatment gives comparison to the experimental group
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Group is given a total of four electroacupuncture treatments to evaluate it's anesthetic effectiveness
  Arms: Electroacupuncture Treatment Group
Device: Sham electroacupuncture — Sham electroacupuncture treatment gives comparison to the experimental group
  Arms: Sham Treatment Group

SUMMARY:
This study is designed to evaluate whether or not electroacupuncture can have an effect on the pain threshold of the subject, as compared to sham treatment.

DETAILED DESCRIPTION:
This study is utilized to evaluate the what effectiveness electroacupuncture has on pain threshold as compared to sham. The outcome measurement utilized will be a digital algometer. The electroacupuncture treatment will consist of a total of four electroacupuncture treatments stimulating acupuncture points LI4 and LI11, and will be given on the same upper extremity tested by the algometer. The algometer measurements will occur alone on the first week, prior to the treatments on the second and third week, and the final reading alone on the fourth week.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy subjects

Exclusion Criteria:

* Hypertension
* Heart Disease
* Pregnancy
* No spinal manipulation or other treatment or medication that could effect pain threshold

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Digital Algometer | Four Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States